CLINICAL TRIAL: NCT03011541
Title: Bone Marrow Derived Stem Cell Ophthalmology Treatment Study II
Brief Title: Stem Cell Ophthalmology Treatment Study II
Acronym: SCOTS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MD Stem Cells (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOTS2
Record Dates: First submitted 2017-01-01; First posted 2017-01-05 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Retinal Disease; Age-Related Macular Degeneration; Retinitis Pigmentosa; Stargardt Disease; Optic Neuropathy; Nonarteritic Ischemic Optic Neuropathy; Optic Atrophy; Optic Nerve Disease; Glaucoma; Leber Hereditary Optic Neuropathy; Blindness; Vision Loss Night; Vision Loss Partial; Vision, Low; Retinopathy; Maculopathy; Macular Degeneration; Retina Atrophy
Keywords: Stem Cells; Bone Marrow Derived Stem Cells; BMSC; Mesenchymal Stem Cells; MSC; Eye Disease; Ophthalmology; Ophthalmic Disease; Retina; Retinal Disease; Macular Degeneration; Age Related Macular Degeneration; Myopic Macular Degeneration; Geographic Atrophy; Dry Macular Degeneration; Wet Macular Degeneration; Retinal Atrophy; Retinal Dystrophy; Hereditary Retinal Dystrophy; Malattia Leventinese; Retinitis Pigmentosa; Stargardt Disease; Cone Dystrophy; Rod-Cone Dystrophy; Cone-Rod Dystrophy; Maculopathy; Optic Nerve Disease; Optic Atrophy; Optic Neuropathy; Ischemic Optic Neuropathy; Optic Nerve Damage; Optic Nerve Compression; Compressive Optic Neuropathy; Devics Syndrome; Ushers Syndrome; Neuromyelitis Optica; Dominant Optic Atrophy; Kjers Optic Atrophy; Leber Hereditary Optic Neuropathy; Blindness; Vision Loss; Retina Atrophy
MeSH Terms: conditions — Retinal Diseases; Macular Degeneration; Retinitis Pigmentosa; Stargardt Disease; Optic Nerve Diseases; Optic Atrophy; Glaucoma; Optic Atrophy, Hereditary, Leber; Blindness; Vitamin A Deficiency; Vision, Low; Eye Diseases; Geographic Atrophy; Wet Macular Degeneration; Retinal Dystrophies; Doyne honeycomb retinal dystrophy; Cone Dystrophy; Cone-Rod Dystrophies; Optic Neuropathy, Ischemic; Optic Nerve Injuries; Neuromyelitis Optica; Usher Syndromes; Optic Atrophy, Autosomal Dominant; Vision Disorders

STUDY DESIGN:
Intervention Model Description: Single Arm- Arm 1. Comparator is natural history of the disease.
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Arm 1 (Other): BMSC provided retrobulbar, subtenon and intravenous for one or both eyes
  Interventions: Procedure: Arm 1

INTERVENTIONS:
Procedure: Arm 1 — Procedure/ Surgery: RB (Retrobulbar)
  Retrobulbar injection of Bone Marrow Derived Stem Cells (BMSC)
  Procedure/Surgery: ST (Subtenon)
  Subtenon injection of Bone Marrow Derived Stem Cells (BMSC)
  Procedure/Surgery: IV (Intravenous)
  Intravenous injection of Bone Marrow Derived Stem Cells (BMSC)
  Other Names: Retrobulbar( RB); Subtenon (ST); Intravenous (IV)

SUMMARY:
This study will evaluate the use of autologous bone marrow derived stem cells (BMSC) for the treatment of retinal and optic nerve damage or disease.

DETAILED DESCRIPTION:
Eyes with loss of vision from retinal or optic nerve conditions generally considered irreversible will be treated with a combination of injections of autologous bone marrow derived stem cells isolated from the bone marrow using standard medical and surgical practices. Retinal conditions may include degenerative, ischemic or physical damage ( examples may include macular degeneration, hereditary retinal dystrophies such as retinitis pigmentosa, stargardt, non-perfusion retinopathies, post retinal detachment. Optic Nerve conditions may include degenerative, ischemic or physical damage ( examples may include optic nerve damage from glaucoma, compression, ischemic optic neuropathy, optic atrophy ). Injections may include retrobulbar, subtenon, intravitreal, intraocular, subretinal and intravenous. Patients will be followed for 12 months with serial comprehensive eye examinations including relevant imaging and diagnostic ophthalmic testing.

ELIGIBILITY:
Inclusion Criteria:

* Have objective, documented damage to the retina or optic nerve unlikely to improve OR
* Have objective, documented damage to the retina or optic nerve that is progressive AND have less than or equal to 20/30 best corrected central visual acuity in one or both eyes AND/OR an abnormal visual field in one or both eyes.
* Be at least 3 months post-surgical treatment intended to treat any ophthalmologic disease and stable.
* If under current medical therapy ( pharmacologic treatment) for a retinal or optic nerve disease be considered stable on that treatment and unlikely to have visual function improvement ( for example, glaucoma with intraocular pressure stable on topical medications but visual field damage ).
* Have the potential for improvement with BMSC treatment and be at minimal risk of any potential harm from the procedure.
* Be over the age of 18
* Be medically stable and able to be medically cleared by their primary care physician or a licensed primary care practitioner for the procedure.
* Medical clearance means that in the estimation of the primary care practitioner, the patient can reasonably be expected to undergo the procedure without significant medical risk to health.

Exclusion Criteria:

* Patients who are not capable of an adequate ophthalmologic examination or evaluation to document the pathology.
* Patients who are not capable or not willing to undergo follow up eye exams with the principle investigator or their ophthalmologist or optometrist as outlined in the protocol.
* Patients who are not capable of providing informed consent.
* Patients who may be at significant risk to general health or to the eyes and visual function should they undergo the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | Change from pre-procedure to 12 months
  Best corrected visual acuity will be measured with Snellen Eye Chart and the ETDRS (Early Treatment Diabetic Retinopathy Study)Eye Chart when available at each post- procedure visit. Intervals at minimum will be first post- procedure day,then 3 months, 6 months and 12 months post-procedure day. Recommended visit 1 month post -procedure day.

SECONDARY OUTCOMES:
Visual Fields | Change from pre-procedure to 12 months
  Visual fields will be evaluated with automated perimetry during post- procedure visits as needed and specifically at 6 months and 12 months. Visual fields are a key measurement in patients with peripheral vision loss.
Optical Coherence Tomography (OCT) | Change from pre-procedure to 12 months
  OCT thickness of the retinal nerve fiber layer the optic nerve and/or macula during the post- procedure visits as needed and specifically at 6 and 12 months - if available.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Levy, MD, Study Chair — MD Stem Cells; Jeffrey Weiss, MD, Principal Investigator — Coral Springs Florida, Vienna Austria, Dubai UAE
Locations (4):
- United States (2):
  - MD Stem Cells, Westport, Connecticut
  - MD Stem Cells, Coral Springs, Florida
- MD Stem Cells Kobinia Med, Vienna, Austria, Austria
- The Saudi-German Hospital, Dubai, United Arab Emirates, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data (IPD)

REFERENCES:
- [Background] Weiss JN, Levy S, Malkin A. Stem Cell Ophthalmology Treatment Study (SCOTS) for retinal and optic nerve diseases: a preliminary report. Neural Regen Res. 2015 Jun;10(6):982-8. doi: 10.4103/1673-5374.158365. PMID 26199618
- [Background] Weiss JN, Levy S, Benes SC. Stem Cell Ophthalmology Treatment Study (SCOTS) for retinal and optic nerve diseases: a case report of improvement in relapsing auto-immune optic neuropathy. Neural Regen Res. 2015 Sep;10(9):1507-15. doi: 10.4103/1673-5374.165525. PMID 26604914
- [Background] Weiss JN, Benes SC, Levy S. Stem Cell Ophthalmology Treatment Study (SCOTS): improvement in serpiginous choroidopathy following autologous bone marrow derived stem cell treatment. Neural Regen Res. 2016 Sep;11(9):1512-1516. doi: 10.4103/1673-5374.191229. PMID 27857759
- [Background] Weiss JN, Levy S, Benes SC. Stem Cell Ophthalmology Treatment Study (SCOTS): bone marrow-derived stem cells in the treatment of Leber's hereditary optic neuropathy. Neural Regen Res. 2016 Oct;11(10):1685-1694. doi: 10.4103/1673-5374.193251. PMID 27904503
- [Background] Weiss JN, Levy S, Benes SC. Stem Cell Ophthalmology Treatment Study: bone marrow derived stem cells in the treatment of non-arteritic ischemic optic neuropathy (NAION). Stem Cell Investig. 2017 Nov 23;4:94. doi: 10.21037/sci.2017.11.05. eCollection 2017. PMID 29270420
- [Background] Weiss JN, Levy S. Stem Cell Ophthalmology Treatment Study: bone marrow derived stem cells in the treatment of Retinitis Pigmentosa. Stem Cell Investig. 2018 Jun 6;5:18. doi: 10.21037/sci.2018.04.02. eCollection 2018. PMID 30050918
- [Background] Weiss JN, Levy S. Dynamic light scattering spectroscopy of the retina-a non-invasive quantitative technique to objectively document visual improvement following ocular stem cell treatment. Stem Cell Investig. 2019 Apr 1;6:8. doi: 10.21037/sci.2019.03.01. eCollection 2019. PMID 31119146
- [Background] Weiss JN, Levy S. Stem Cell Ophthalmology Treatment Study (SCOTS): bone marrow derived stem cells in the treatment of Usher syndrome. Stem Cell Investig. 2019 Sep 9;6:31. doi: 10.21037/sci.2019.08.07. eCollection 2019. PMID 31620478
- [Background] Weiss JN, Levy S. Stem Cell Ophthalmology Treatment Study (SCOTS): bone marrow derived stem cells in the treatment of Dominant Optic Atrophy. Stem Cell Investig. 2019 Dec 5;6:41. doi: 10.21037/sci.2019.11.01. eCollection 2019. PMID 32039263
- [Background] Weiss JN, Levy S. Stem Cell Ophthalmology Treatment Study (SCOTS): Bone Marrow-Derived Stem Cells in the Treatment of Age-Related Macular Degeneration. Medicines (Basel). 2020 Mar 28;7(4):16. doi: 10.3390/medicines7040016. PMID 32231088
- [Background] Weiss JN, Levy S. Stem Cell Ophthalmology Treatment Study (SCOTS): Bone Marrow-Derived Stem Cells in the Treatment of Stargardt Disease. Medicines (Basel). 2021 Feb 3;8(2):10. doi: 10.3390/medicines8020010. PMID 33546345